CLINICAL TRIAL: NCT00662090
Title: Prospective Non-randomized Multi-center Study for Epidemiology and Characterization of Myelodysplastic Syndromes (MDS) and Juvenile Myelomonocytic Leucemia (JMML) in Childhood
Brief Title: Study for Epidemiology and Characterization of Myelodysplastic Syndromes (MDS) and Juvenile Myelomonocytic Leucemia (JMML) in Childhood
Acronym: EWOG MDS 2006
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Charlotte Niemeyer, MD, Prof. Dr. Charlotte Niemeyer, MD, University Hospital Freiburg
Other Study IDs: EWOG MDS 2006; NCT00898339 (obsolete NCT alias)
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Myelodysplastic Syndromes; Juvenile Myelomonocytic Leukemia
Keywords: MDS; JMML; EWOG-MDS; Myelodysplastic Syndromes (MDS); Juvenile Myelomonocytic Leukemia (JMML)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Juvenile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At diagnosis, prior to HSCT and at relapse material form peripheral blood and bone marrow will be retrieved and stored for research purposes. If there are other diagnostic bone marrow examinations at other time points (prior to HSCT), the material will be handled the same way.
  The following material will be retrieved:
  * 8 smears from PB
  * 8 smears from BM
  * at least 5 ml of heparinized PB
  * at least 5 ml of heparinized BM
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to improve the accuracy of diagnosis for children and adolescents with MDS by a standardized review of morphology and standardized cytogenetic and molecular analysis.

The primary objectives of the study are:

* To evaluate the frequency of the different subtypes of MDS in childhood and adolescence by a standardized diagnostic approach
* To evaluate the frequency of cytogenetic and molecular abnormalities:

Specifically using array-CGH to evaluate the frequency of subtle chromosomal imbalances, i.e. gains and losses of defined chromosomal regions, and amplifications.

Specifically using mFISH to identify unknown chromosomal aberrations, particularly subtle translocations involving new candidate genes, and to better define chromosomal breakpoints.

The secondary objectives of the study are:

* To assess survival for children and adolescents with MDS and JMML
* To evaluate relapse rate, morbidity and mortality in children with MDS and JMML treated by HSCT

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by the caretakers and whenever possible the patient's assent.
* Confirmed diagnosis of MDS or JMML (morphology, cytogenetics)
* Myeloid leukemia of Down syndrome (patients aged > 6 years).
* Age less than 18 years

Exclusion Criteria:

* Denied informed consent and/or assent by caretakers/patient.
* Myeloid leukemia of Down syndrome (patients < 6 years).
* Participation in another study within the last 4 weeks (except for therapy optimizing studies in cancer or bone marrow failure disorders and studies in diagnostics).

Max Age: 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: MDS and JMML diagnosted
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2006-01; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the frequency of the different subtypes of MDS in childhood and adolescence by a standardized diagnostic approach | 5 years
To evaluate the frequency of cytogenetic and molecular abnormalities | 5 years

SECONDARY OUTCOMES:
To assess survival for children and adolescents with MDS and JMML | 5 years
To evaluate relapse rate, morbidity and mortality in children with MDS and JMML treated by HSCT | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte M. Niemeyer, M.D., Principal Investigator — University of Freiburg
Locations (1):
- University Hospital of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Drexler B, Schwarz-Furlan S, Baumann I, Rudelius M, Nollke P, Lebrecht D, Ramamoorthy S, Rotari N, Karow A, Hirabayashi S, Beier F, Behrens YL, Gohring G, Kalb R, Wlodarski MW, Strahm B, Erlacher M, Niemeyer CM, Yoshimi A. Long-term outcomes of patients with refractory cytopenia of childhood under observation only. Blood Adv. 2025 Aug 26;9(16):4279-4285. doi: 10.1182/bloodadvances.2025016136. PMID 40554414
- [Derived] Erlacher M, Andresen F, Sukova M, Stary J, De Moerloose B, Bosch JVWT, Dworzak M, Seidel MG, Polychronopoulou S, Beier R, Kratz CP, Nathrath M, Fruhwald MC, Gohring G, Bergmann AK, Mayerhofer C, Lebrecht D, Ramamoorthy S, Yoshimi A, Strahm B, Wlodarski MW, Niemeyer CM. Spontaneous remission and loss of monosomy 7: a window of opportunity for young children with SAMD9L syndrome. Haematologica. 2024 Feb 1;109(2):422-430. doi: 10.3324/haematol.2023.283591. PMID 37584291
- [Derived] Jorgensen SF, Buechner J, Myhre AE, Galteland E, Spetalen S, Kulseth MA, Sorte HS, Holla OL, Lundman E, Alme C, Heier I, Flaegstad T, Floisand Y, Benneche A, Fevang B, Aukrust P, Stray-Pedersen A, Gedde-Dahl T, Nordoy I. A Nationwide Study of GATA2 Deficiency in Norway-the Majority of Patients Have Undergone Allo-HSCT. J Clin Immunol. 2022 Feb;42(2):404-420. doi: 10.1007/s10875-021-01189-y. Epub 2021 Dec 10. PMID 34893945
- [Derived] Aalbers AM, van den Heuvel-Eibrink MM, Baumann I, Dworzak M, Hasle H, Locatelli F, De Moerloose B, Schmugge M, Mejstrikova E, Novakova M, Zecca M, Zwaan CM, Te Marvelde JG, Langerak AW, van Dongen JJ, Pieters R, Niemeyer CM, van der Velden VH. Bone marrow immunophenotyping by flow cytometry in refractory cytopenia of childhood. Haematologica. 2015 Mar;100(3):315-23. doi: 10.3324/haematol.2014.107706. Epub 2014 Nov 25. PMID 25425683
- [Derived] Aalbers AM, van den Heuvel-Eibrink MM, Baumann I, Beverloo HB, Driessen GJ, Dworzak M, Fischer A, Gohring G, Hasle H, Locatelli F, De Moerloose B, Noellke P, Schmugge M, Stary J, Yoshimi A, Zecca M, Zwaan CM, van Dongen JJ, Pieters R, Niemeyer CM, van der Velden VH, Langerak AW. T-cell receptor Vbeta skewing frequently occurs in refractory cytopenia of childhood and is associated with an expansion of effector cytotoxic T cells: a prospective study by EWOG-MDS. Blood Cancer J. 2014 May 2;4(5):e209. doi: 10.1038/bcj.2014.28. PMID 24786393
- [Derived] Yoshimi A, van den Heuvel-Eibrink MM, Baumann I, Schwarz S, Simonitsch-Klupp I, de Paepe P, Campr V, Kerndrup GB, O'Sullivan M, Devito R, Leguit R, Hernandez M, Dworzak M, de Moerloose B, Stary J, Hasle H, Smith OP, Zecca M, Catala A, Schmugge M, Locatelli F, Fuhrer M, Fischer A, Guderle A, Nollke P, Strahm B, Niemeyer CM. Comparison of horse and rabbit antithymocyte globulin in immunosuppressive therapy for refractory cytopenia of childhood. Haematologica. 2014 Apr;99(4):656-63. doi: 10.3324/haematol.2013.095786. Epub 2013 Oct 25. PMID 24162791
- [Derived] Gohring G, Michalova K, Beverloo HB, Betts D, Harbott J, Haas OA, Kerndrup G, Sainati L, Bergstraesser E, Hasle H, Stary J, Trebo M, van den Heuvel-Eibrink MM, Zecca M, van Wering ER, Fischer A, Noellke P, Strahm B, Locatelli F, Niemeyer CM, Schlegelberger B. Complex karyotype newly defined: the strongest prognostic factor in advanced childhood myelodysplastic syndrome. Blood. 2010 Nov 11;116(19):3766-9. doi: 10.1182/blood-2010-04-280313. Epub 2010 Aug 27. PMID 20802024
- See also: Homepage of the EWOG-MDS-Study Group — http://www.ewog-mds.org